CLINICAL TRIAL: NCT00089102
Title: Phase II Study of Gemcitabine and CPT-11 (Irinotecan) in Unresectable or Metastatic Renal Cell Carcinoma
Brief Title: Gemcitabine and Irinotecan in Treating Patients With Locally Advanced Unresectable or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000378044; MUSC-100730; MUSC-HR-10981; PHARMACIA-B9E-US-X388; LILLY-MUSC-100730
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine + Irinotecan (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 1,000 mg/m2/dose in 250 cc of NS IV over 30 minutes on Days 1 and 8 of each 21 day cycle
Drug: irinotecan hydrochloride — 100mg/m2/dose in 500 cc of D5W or NS IV over 90 minutes on days 1 and 8 of each 21 day cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and irinotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with irinotecan works in treating patients with locally advanced unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine response in patients with locally advanced unresectable or metastatic renal cell carcinoma treated with gemcitabine and irinotecan.

Secondary

* Determine the duration of response in patients treated with this regimen.
* Determine the tolerance to and toxicity of this regimen in these patients.
* Determine median and progression-free survival in patients treated with this regimen.

OUTLINE: Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for 6-8 courses in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses beyond best response.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 12-36 patients will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Locally advanced unresectable or metastatic disease
* Unidimensionally measurable disease by physical exam or imaging study

  * The following are not considered measurable disease:

    * Bone only disease
    * Pleural or peritoneal effusions
    * CNS lesions
    * Irradiated lesions unless disease progression was documented after radiotherapy

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* ALT and AST < 3 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL

Gastrointestinal

* No active inflammatory bowel disease
* No significant bowel obstruction
* No chronic diarrhea

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No mental incapacitation or psychiatric illness that would preclude giving informed consent
* No other active malignancy except nonmelanoma skin cancer
* No other severe disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormones except steroids for adrenal failure, hormones for non-disease-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery

* Not specified

Other

* No concurrent participation in another clinical trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uzair B. Chaudhary, MD, Principal Investigator — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (2):
- United States (2):
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + Irinotecan
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Irinotecan
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Proportion
Time Frame: From registration until time of complete response or partial response
Population: All patients treated on study who underwent a response assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + Irinotecan
Number analyzed (Participants) | 7
Participants
  Complete response | 1
  Partial Response | 4
  Stable or Progressive Disease | 2

2. Secondary Outcome: Duration of Response
Time Frame: From registration until disease progression among patients who had at least a partial response
Population: Data is not available for this endpoint was not collected.
Arm/Group | Gemcitabine + Irinotecan
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Who Experienced SAEs on Study
Time Frame: From the day of first dose until the end of study, for an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + Irinotecan
Number analyzed (Participants) | 9
Participants
  Number of patients who experienced an SAE | 4
  Number of patients who did not experience an SAE | 5

4. Secondary Outcome: Progression-free Survival
Time Frame: Time between registration and disease progression or death, whichever comes first.
Population: Data for this endpoint was not collected
Arm/Group | Gemcitabine + Irinotecan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From day 1 until end of study visit, an average of 6 months
Description: Data for adverse events (non-serious) was not collected.
Arm/Group | Gemcitabine + Irinotecan
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Irinotecan (N=9)
left pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cerebrovascular accident (General disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes